CLINICAL TRIAL: NCT01608373
Title: Comparison of Intravenous Lidocaine and Intraperitoneal Lidocaine Irrigation for Effective Pain Relief After Laparoscopic Cholecystectomy: A Prospective, Randomized, Double-blind, Placebo-controlled Study
Brief Title: The Effect of Intravenous Lidocaine and Intraperitoneal Lidocaine Irrigation on Pain After Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, Hyun Kang, Assistant professor, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChungAngUH4
Record Dates: First submitted 2012-05-26; First posted 2012-05-31 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2011-07

CONDITIONS: Postoperative Pain
Keywords: Pain; Lidocaine; Intravenous; Intraperitoneum; Laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intravenous lidocaine injection group (Active Comparator): Patients in Group I (intravenous lidocaine injection group) received an intravenous bolus injection of 1.5 mg/kg lidocaine followed by a continuous lidocaine infusion of 2 mg/kg/hr.
  Interventions: Drug: Intravenous lidocaine injection
- Intraperitoneal lidocaine irrigation group (Active Comparator): Patients in Group P(intraperitoneal lidocaine irrigation group) receive a peritoneal lidocaine irrigation with 3.5mg/kg lidocaine and normal saline 100cc.
  Interventions: Drug: Intraperitoneal lidocaine irrigation group
- Intravenous normal saline group (Placebo Comparator): The patients in Group C (placebo control group) received normal saline intravenous injection
  Interventions: Drug: Intravenous normal saline injection

INTERVENTIONS:
Drug: Intravenous lidocaine injection — Patients in Group I (intravenous lidocaine injection group) received an intravenous bolus injection of 1.5 mg/kg lidocaine followed by a continuous lidocaine infusion of 2 mg/kg/hr
  Other Names: IV lidocaine
  Arms: Intravenous lidocaine injection group
Drug: Intraperitoneal lidocaine irrigation group — Patients in Group P(intraperitoneal lidocaine irrigation group) receive a peritoneal lidocaine irrigation with 3.5mg/kg lidocaine and normal saline 100cc. 50cc of irrigation fluid will be spread below diaphragm and 50cc of irrigation fluid will be spread around the gall bladder.
  Other Names: IP lidocaine
  Arms: Intraperitoneal lidocaine irrigation group
Drug: Intravenous normal saline injection — The patients in Group C (placebo control group) received normal saline intravenous injection
  Other Names: IV normal saline
  Arms: Intravenous normal saline group

SUMMARY:
This prospective randomized study aims to comparison the effectiveness of intravenous lidocaine injection and intraperitoneam lidocaine irrigation on the relief of pain in patients undergoing laparoscopic cholecystectomy.

A total of 83 patients will be randomized into one of three groups (group C or group I or group P) based on Excel number generation.

Patients in group C will receive normal saline intravenous injection, and patients in group I will receive an intravenous bolus injection of 1.5 mg/kg lidocaine followed by a continuous lidocaine infusion of 2 mg/kg/hr.

Patients in group P will receive intraperitoneal lidocaine irrigation with 3.5 mg/kg lidocaine and normal saline 100cc.

Visual analogue scale pain scores, fentanyl consumption and the frequency at which patients pushed the button (FPB) of a patient-controlled analgesia system will be recorded at 2, 4, 8, 12, 24, 48 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic cholecystectomy

Exclusion Criteria:

* mental change
* allergy to local anesthetics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain measuring using Visual analogue scale at postoperative 2hour | Post op 2 hour
  Patients will be assessed for pain using a visual analogue pain scale (VAS). It is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 2hour.

SECONDARY OUTCOMES:
Visual analogue scale 4hour | Post op 4 hour
  Patients will be assessed for pain using a visual analogue pain scale (VAS). It is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 4hour.
Visual analogue scale 8hour | Post op 8 hour
  Patients will be assessed for pain using a visual analogue pain scale (VAS). It is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 8hour.
Visual analogue scale 12 hour | Post op 12hour
  Patients will be assessed for pain using a visual analogue pain scale (VAS). It is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 12hour.
visual analogue scale 24hour | Post op 24hour
  Patients will be assessed for pain using a visual analogue pain scale (VAS). It is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 24hour.
Visual analogue scale 48 hour | Post op 48hour
  Patients will be assessed for pain using a visual analogue pain scale (VAS). It is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 48hour.
Opioid consumption 2hour | Post op 2 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. In the case of persistent pain greater than a visual analogue scale (VAS) pain score of 30 mm, an additional 50 μg of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30 mm. And sum of delivery from PCA system and additional opioid fom immediately after operation to post op 2hour will be measured.
Opioid consumption 4 hour | Post op 4 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. In the case of persistent pain greater than a visual analogue scale (VAS) pain score of 30 mm, an additional 50 μg of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30 mm. And sum of delivery from PCA system and additional opioid fom immediately after operation to post op 4hour will be measured.
Opioid consumption 8 hour | Post op 8 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. In the case of persistent pain greater than a visual analogue scale (VAS) pain score of 30 mm, an additional 50 μg of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30 mm. And sum of delivery from PCA system and additional opioid fom immediately after operation to post op 8hour will be measured.
Opioid consumption 12 hout | Post op 12 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. In the case of persistent pain greater than a visual analogue scale (VAS) pain score of 30 mm, an additional 50 μg of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30 mm. And sum of delivery from PCA system and additional opioid fom immediately after operation to post op 12hour will be measured.
Opioid consumption 24 hour | Post op 24 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. In the case of persistent pain greater than a visual analogue scale (VAS) pain score of 30 mm, an additional 50 μg of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30 mm. And sum of delivery from PCA system and additional opioid fom immediately after operation to post op 24hour will be measured.
Opioid consumption 48hour | Post op 48 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. In the case of persistent pain greater than a visual analogue scale (VAS) pain score of 30 mm, an additional 50 μg of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30 mm. And sum of delivery from PCA system and additional opioid fom immediately after operation to post op 48hour will be measured.
FPB 2 hour | Post op 2 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And total frequency of patient to push the button of the PCA machine (FPB) fom immediately after operation to post op 2 hour will be measured.
FPB 4 hour | Post op 4 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And total frequency of patient to push the button of the PCA machine (FPB) fom immediately after operation to post op 4 hour will be measured.
FPB 8 hour | Post op 8 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And total frequency of patient to push the button of the PCA machine (FPB) fom immediately after operation to post op 8 hour will be measured.
FPB 12 hour | Post op 12 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And total frequency of patient to push the button of the PCA machine (FPB) fom immediately after operation to post op 12 hour will be measured.
FPB 24 hour | Post op 24hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And total frequency of patient to push the button of the PCA machine (FPB) fom immediately after operation to post op 24 hour will be measured.
FPB 48 hour | Post op 48 hour
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And total frequency of patient to push the button of the PCA machine (FPB) fom immediately after operation to post op 48 hour will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Kang, Ph.D, Study Chair — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Eun Jin Ahn, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Hyun Kang, Seoul, South Korea

REFERENCES:
- [Derived] Yang SY, Kang H, Choi GJ, Shin HY, Baek CW, Jung YH, Choi YS. Efficacy of intraperitoneal and intravenous lidocaine on pain relief after laparoscopic cholecystectomy. J Int Med Res. 2014 Apr;42(2):307-19. doi: 10.1177/0300060513505493. PMID 24648482